CLINICAL TRIAL: NCT05282342
Title: Comparative Analysis of the Health Status of Heart Transplant Patients With Different Levels of Physical Activity
Brief Title: Heart Transplant Patients, Health Status and Physical Activity
Status: Completed | Type: Observational
Sponsor: Luis Santos (Other)
Responsible Party: Sponsor-Investigator, Luis Santos, Sponsor-Investigator, University of Oviedo
Organization: University of Oviedo (Other)
Other Study IDs: ETICA-ULE-038-2021
Record Dates: First submitted 2021-12-29; First posted 2022-03-16 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Disease, Chronic
MeSH Terms: conditions — Chronic Disease | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Transplanted with low levels of physical activity (TPL)
  Interventions: Diagnostic Test: Diagnostic tests
- Transplanted with moderate levels of physical activity (TPM)
  Interventions: Diagnostic Test: Diagnostic tests
- Transplanted with high levels of physical activity (TPH)
  Interventions: Diagnostic Test: Diagnostic tests
- Healthy sedentary individuals (S)
  Interventions: Diagnostic Test: Diagnostic tests

INTERVENTIONS:
Diagnostic Test: Diagnostic tests — No intervention will be carried out. Participants of the whole groups will be underwent the same tests.

SUMMARY:
The aim of this cross-sectional observational study is (1) to assess the health status of a group of heart transplant patients and their level of physical activity, (2) and to compare the health status of a group of heart transplant patients with different levels of physical activity, with a group of healthy people classified as sedentary (due to their level of physical activity).

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant adults (18 years old) whose transplant had taken place at least twelve months before the study data was taken.
* Heart transplant patients with low, moderate and high levels of physical activity, according to the results of the International Physical Activity Questionnaire - Long Form (IPAQ-L).
* Healthy people with low levels of physical activity, according to the results of the International Physical Activity Questionnaire - Long Form (IPAQ-L).

Exclusion Criteria:

* Do not meet the eligibility criteria.
* Have physical disabilities and/or other limiting pathologies that would condition their level of physical activity.
* Have participated in cardiac rehabilitation programs during the twelve months prior to the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active and sedentary heart transplant patients and sedentary healthy people.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Cardiovascular function assessment. | Through study completion, an average of 1 year.
  Analysis of several cardiovascular variables.
Neuromuscular function assessment. | through study completion, an average of 1 year
  Analysis of several neuromuscular variables.

SECONDARY OUTCOMES:
Basic blood analysis | Through study completion, an average of 1 year.
  Analysis of several blood parameters
Flexibility | Through study completion, an average of 1 year.
  Analysis of several flexibility variables.
Balance | Through study completion, an average of 1 year.
  Analysis of several balance variables.
Functional Capacity | Through study completion, an average of 1 year.
  Analysis of several functional mobility variables.
Quality of Life Status | Through study completion, an average of 1 year.
  Analysis of several quality of life variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Itziar Salas Reguera, León, León, Castilla Y León, Spain